CLINICAL TRIAL: NCT06091007
Title: The Effects of Magnesium Citrate Supplementation on Hand Grip Strength: A Randomized Control Trial
Brief Title: Magnesium Citrate Supplementation on Hand Grip Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5230401
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Hand Grasp
Keywords: hand grip magnesium citrate
MeSH Terms: interventions — Magnesium

STUDY DESIGN:
Intervention Model Description: Group 1: participants take 200 mg of magnesium citrate daily for 4 weeks. Group 2: participants take 400 mg of magnesium citrate daily for 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 200 mg Magnesium (Active Comparator): Participant will take 200 mg of magnesium citrate daily for 4 weeks
  Interventions: Dietary Supplement: Magnesium
- 400 mg Magnesium (Active Comparator): Participant will take 400 mg of magnesium citrate daily for 4 weeks
  Interventions: Dietary Supplement: Magnesium

INTERVENTIONS:
Dietary Supplement: Magnesium — Magnesium citrate of either 200mg or 400 mg will be taken by the participant with food in the morning.

SUMMARY:
The purpose of this research study is to determine the effectiveness of magnesium on handgrip strength using the more bioavailable magnesium citrate.

DETAILED DESCRIPTION:
In this single-blind, randomized trial, participants will take a daily dose of either 200 or 400 milligrams of magnesium citrate supplement for four weeks, perform three separate handgrip strength tests using a dynamometer, complete a demographics questionnaire, a physical activity questionnaire, and a compliance log.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy community adults
* Individuals age 18 and over
* Male and female participants

Exclusion Criteria:

* Individuals currently on magnesium supplements
* Individuals currently on a multivitamin supplement
* Individuals who currently suffer from hand pain or hand injury
* Individuals who currently suffer from arthritis in their hands
* Individuals suffering from a gastrointestinal disorder complicated by diarrhea, nausea, or abdominal cramping

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | change between baseline and 4 weeks
  Participants will perform three separate handgrip strength tests using a Jamar Plus digital hand dynamometer, (Sammons Preston, Bolingbrook, Illinois).
  In each test, participants will do three trials resting for 15 seconds between trials, the average of the three trials will be recorded. To perform the hand grip strength test, the participant will hold the dynamometer in their dominant hand, with the arm at a right angle, and with the elbow by the side of the body. The participant then squeezes the hand dynamometer with maximum isometric effort for at least five seconds. Participants are required to not move any other part of the body and are encouraged to use maximum effort.

CONTACTS AND LOCATIONS:
Overall Officials: Kyndra Woosley, MS, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States